CLINICAL TRIAL: NCT00004912
Title: Phase II Trial of Progressive Resistance Training With Megestrol Acetate for the Treatment of Cancer-Related Weight Loss
Brief Title: Megestrol and Exercise in Treating Patients With Cancer-Related Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: NU FDA98CC6; NU-98CC6; NCI-G00-1705
Record Dates: First submitted 2000-03-07; First posted 2004-03-03 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cachexia; Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; fatigue; cachexia
MeSH Terms: conditions — Cachexia; Fatigue | interventions — Megestrol Acetate; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: megestrol acetate
Procedure: physical therapy

SUMMARY:
RATIONALE: Megestrol helps improve appetite. Exercise may decrease cancer-related fatigue, improve strength, and build up lost muscle tissue. Exercise plus megestrol may be effective treatment for cancer-related weight loss.

PURPOSE: Phase II trial to study the effectiveness of megestrol plus exercise to improve appetite, increase strength, gain lean body tissue, and decrease fatigue in patients who have cancer-related weight loss.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of megestrol and progressive resistance training on lean body mass, total body weight, functional capacity, appetite, and fatigue in patients with weight loss due to advanced malignancy.

OUTLINE: This is a multicenter study. Patients receive oral megestrol once daily. Patients also begin progressive resistance training 3 days a week. Treatment/exercise continues for 12 weeks in the absence of unacceptable toxicity or progressive weight loss (greater than 5 pounds or 5% or more over first 4 study weeks).

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Advanced nonhormone responsive malignancy (metastatic or incurable) Nonvolitional weight loss of between 6-9% of usual body weight over past 6 months OR Decrease of 5 pounds in the past 2 months or less (not greater than 10% loss of usual body weight) No clinical or radiologic evidence of ascites or pleural effusion No lytic bone metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-1 Life expectancy: At least 4 months Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No venous thrombosis No congestive heart failure Other: Able to participate in exercise program for 1 hour, 3 times/week No physical handicap that precludes aerobic or resistance exercise No clinical abnormality that renders exercise a risk At least 1 month since strength training of 3 hours or more per week No physical or functional obstruction to food intake No uncontrolled emesis greater than 5 episodes/week No diarrhea greater than 4 stools/day intractable to antidiarrheal medication No IV hyperalimentation No contraindications to megestrol No dementia or mental incompetence No known AIDS Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: No concurrent adrenal steroids (other than for replacement), anabolics, appetite stimulants, or progestational agents Intermittent corticosteroids as antiemetic or premedication for cancer treatment allowed At least 6 weeks since prior megestrol Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hayden Von Roenn, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (6):
- United States (6):
  - University of Arkansas - Department of Geriatrics, North Little Rock, Arkansas
  - Pacific Shores Medical Group, Long Beach, California
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Office of David Cella, Evanston, Illinois
  - Rex Healthcare, Raleigh, North Carolina